CLINICAL TRIAL: NCT00518037
Title: Quality of Life in Patients With Nonmelanoma Skin Cancer
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery and Surgery-Organ Transplantation, Northwestern University
Other Study IDs: 1253-006
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Nonmelanoma Skin Cancer
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: nonmelanoma skin cancer patients
  Interventions: Behavioral: surveys

INTERVENTIONS:
Behavioral: surveys — anxiety surveys

SUMMARY:
The goal of this study is to learn more about the physical discomfort, sensory impairment, depression, anxiety, and interference with relationships, family, and work associated with NMSC via survey questions.

DETAILED DESCRIPTION:
The purpose of this study is to learn more about the physical discomfort, sensory impairment, depression, anxiety, and interference with relationships, family, and work associated with NMSC via survey questions.

ELIGIBILITY:
Inclusion Criteria:

* patients with nonmelanoma skin cancer
* 18 years of age

Exclusion Criteria:

* non-English speakers
* minors

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: nonmelanoma skin cancer patients
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2006-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
statistics from results of Skindex survey | 1 hour to complete survey

SECONDARY OUTCOMES:
statistics from time-tradeoff utility survey | 1 hour to complete survey

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern University Dermatology, Chicago, Illinois